CLINICAL TRIAL: NCT01360580
Title: Current Care Study of Incidence and Consequences of Swallowing Disorders After Invasive Mechanical Ventilation
Brief Title: Swallowing Disorders After Prolonged Mechanical Ventilation
Acronym: Deglutube
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/110/HP; 2008-A00057-50 (Other: Id RCB)
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Larynx Disease
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Epidemiology study for evaluation of incidence of swallowing disorders (SD) after prolonged invasive ventilation (more than seven days), using a clinical statement. All consecutive patients are screened, and clinical evaluation is performed during 48h after patient's extubation. If a SD exist, a new evaluation is realized 48h after. Three groups will be created (1.no SD, 2.transitory SD and 3.persistent SD (eg persistent after 48h)). Data complementary are notified at day 28 (pneumonia? nutritional status?)

ELIGIBILITY:
Inclusion Criteria:

* More than 7 days of invasive mechanical ventilation

Exclusion Criteria:

* Age < 18 years old
* Preexistent swallowing disorders, stroke, tracheostomy
* Failure of patient's agreement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: More than 7d of invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of swallowing disorders after prolonged invasive ventilation | 48 hours after extubation

SECONDARY OUTCOMES:
Nutritional status at day 28 | day 28

CONTACTS AND LOCATIONS:
Overall Officials: Gaetan Beduneau, Doctor, Principal Investigator — Service de Réanimation médicale Hôpitaux de Rouen
Locations (2):
- France (2):
  - Service de Réanimation Médicale, Angers
  - service de Réanimation médicale, Rouen

REFERENCES:
- [Derived] Beduneau G, Souday V, Richard JC, Hamel JF, Carpentier D, Chretien JM, Bouchetemble P, Laccoureye L, Astier A, Tanguy V, Mercat A, Beloncle F, Tamion F. Persistent swallowing disorders after extubation in mechanically ventilated patients in ICU: a two-center prospective study. Ann Intensive Care. 2020 Oct 14;10(1):138. doi: 10.1186/s13613-020-00752-x. PMID 33052476